CLINICAL TRIAL: NCT06000514
Title: Association of Topical Sm29 in Gold Nanoparticles With Intravenous Meglumine Antimoniate in the Treatment of Cutaneous Leishmaniasis Caused by Leishmania Braziliensis: A Randomized Controlled Trial.
Brief Title: Topical Sm29 in Combination With Meglumine Antimoniate in the Treatment of Cutaneous Leishmaniasis.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Paulo Roberto Lima Machado, Head of Immunology Service, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM29CL.1
Record Dates: First submitted 2023-07-19; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cutaneous Leishmaniasis, American
Keywords: Cutaneous Leishmaniasis; Sm29; L. braziliensis
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Leishmaniasis, Cutaneous | interventions — Sm29 protein, Schistosoma mansoni

STUDY DESIGN:
Intervention Model Description: Randomized and controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Both arms will use the same active standard medication (Sbv) and both arms will use a topical cream (one arm - placebo; the other Sm29).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Sm29 and Sbv (Experimental): Use of topical Sm29 twice a day during 20 days and systemic Sbv during 20 days
  Interventions: Drug: Sm29 Protein, Schistosoma Mansoni; Drug: Pentavalent antimony (Sbv)
- Topical Placebo and Sbv (Placebo Comparator): Use of topical placebo twice a day during 20 days and systemic Sbv during 20 days
  Interventions: Drug: Pentavalent antimony (Sbv)

INTERVENTIONS:
Drug: Sm29 Protein, Schistosoma Mansoni — Sm29 cream twice a day in the ulcer(s), during 20 days; and Systemic IV Pentavalent antimony (Sbv) at 20mg/kg/day during 20 days.
  Other Names: Pentavalent antimony (Sbv)
  Arms: Topical Sm29 and Sbv
Drug: Pentavalent antimony (Sbv) — Placebo cream twice a day in the ulcer(s), during 20 days; and Systemic IV Pentavalent antimony (Sbv) at 20mg/kg/day during 20 days.
  Other Names: Placebo cream

SUMMARY:
This project is composed of a phase I study with the purpose of evaluating adverse reactions and the best dose to be used of Sm29 and a phase II randomized controlled study with 3 arms with the purpose of comparing the efficacy of meglumine antimoniate associated with Sm29, with meglumine antimoniate plus placebo and meglumine antimoniate alone in the treatment of cutaneous leishmaniasis.

DETAILED DESCRIPTION:
The phase I study was performed in 10 healthy subjects and 10 patients with CL. In healthy individuals (N=5) Sm29 was applied to healthy skin at a concentration of 5ug and in another 5 Sm29 was used at a dose of 10ug applied twice a day for 20 days. A phase I study was also carried out in 10 patients with CL to assess the occurrence of adverse reactions to Sm29 applied to the ulcerated lesion and to compare the use of two doses of Sm29. In 5 patients, Sm29 was used at a dose of 5ug and applied twice a day, and in 10 patients, a dose of 10ug of Sm29 was used, also applied twice a day. The 10 patients were also treated with glucantime at a dose of 20mg/kg/weight with a maximum dose of 1200mg/day intravenously for 20 days. Patients were evaluated on days 10, 20 and 30 for adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of cutaneous leishmaniasis (typical ulcerated lesion); 1 to 2 ulcers; ulcer size ranging from 10-40mm; disease duration between 20-90 days.

Exclusion Criteria:

* Diabetes; Cardiovascular or kidney disease; HIV seropositivity; use of immunosupressive drugs; pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Cure | 90 days
  Complete re epithelization of the ulcer(s), without any area of ulceration and without raised or infiltrated borders.

CONTACTS AND LOCATIONS:
Overall Officials: SERGIO C OLIVEIRA, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Corte de Pedra Health Post, Presidente Tancredo Neves, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No
Not to be shared.

REFERENCES:
- [Derived] Lago T, Peixoto F, Mambelli F, Carvalho LP, Guimaraes LH, Carvalho AM, Cardoso L, Machado PRL, Scott P, Lago J, Andrade JM, Fahel JS, Oliveira SC, Carvalho EM. Use of topical rSm29 in combination with intravenous meglumine antimoniate in the treatment of cutaneous leishmaniasis: A randomized controlled trial. Int J Infect Dis. 2024 Oct;147:107206. doi: 10.1016/j.ijid.2024.107206. Epub 2024 Aug 13. PMID 39147194